CLINICAL TRIAL: NCT01884935
Title: A Phase 1, Multicenter, Open-Label, Single-Arm, Multiple Dose Study to Evaluate the the Pharmacokinetics and Pharmacodynamics of Natalizumab in Pediatric Subjects With Relapsing Remitting Multiple Sclerosis (RMS)
Brief Title: PK and PD Study of Natalizumab in Pediatric Subjects With RRMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MS328; 2012-005082-13
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2015-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Pediatric
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab (Experimental): 300 mg intravenously (IV) every 4 weeks
  Interventions: Biological: Natalizumab

INTERVENTIONS:
Biological: Natalizumab — As specified in the treatment arm
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective of the study is to determine the pharmacokinetic (PK) profile of multiple doses of natalizumab in pediatric subjects with relapsing-remitting multiple sclerosis (RRMS). The secondary objectives are as follows: to characterize the pharmacodynamic (PD) profile of natalizumab (as defined by α4 integrin binding) and to explore the safety and tolerability of multiple doses of natalizumab in the pediatric population.

ELIGIBILITY:
Key Inclusion Criteria:

- Rapidly evolving severe relapsing remitting multiple sclerosis, defined by 2 or more disabling relapses in 1 year, and with 1 or more gadolinium-enhancing lesions on brain MRI or a significant increase in T2 lesion load, as compared to a previous recent magnetic resonance imaging (MRI)

Key Exclusion Criteria:

* History of, or abnormal laboratory values indicative of, significant medical, neurologic (other than MS), or psychiatric disorders that might preclude participation in the study in the opinion of the Investigator.
* Prior natalizumab therapy.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
predose (trough) concentrations from multiple dosing (Cpredose) | Up to week 16
maximum plasma concentration (Cmax) | Up to Week 16
time to maximum plasma concentration (Tmax) | Up to Week 16
area under the plasma concentration curve from time of first dose to infinity (AUCinf) | Up to Week 16
apparent clearance (Cl/F) | Up to Week 16
volume of distribution | Up to Week 16
elimination half-life (t1/2) | Up to Week 16

SECONDARY OUTCOMES:
the average and minimum saturation values of α4 integrin over the dosing interval | Up to Week 16
incidence of serious adverse events (SAEs), infusion and hypersensitivity reactions, and other AEs | Up to Week 16
the presence of anti-natalizumab antibodies | Up to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- Italy (5):
  - Research Site, Cefalù
  - Research Site, Gallarate
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Rome

REFERENCES:
- See also: EudraCT Tabulated Result — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-005082-13/results